CLINICAL TRIAL: NCT03587974
Title: Cluster Randomized Controlled Trial to Test the Feasibility, Acceptability and Preliminary Effectiveness of a Psychosocial Intervention to Support Alzheimer's Family Caregivers in Vietnam
Brief Title: Randomized Controlled Trial to Test an Alzheimer's Family Caregiver Intervention in Vietnam
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 1223433
Record Dates: First submitted 2018-07-03; First posted 2018-07-16 (Actual); Results first posted 2020-07-22 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Family Caregivers

STUDY DESIGN:
Intervention Model Description: Cluster randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REACH-VN (Experimental): In-home psychosocial intervention to enhance caregiver knowledge and skills and to reduce stress delivered in 4-6 sessions over the course of 2-3 months
  Interventions: Behavioral: REACH-VIETNAM
- Enhanced control (No Intervention): Single session with education about nature of dementia

INTERVENTIONS:
Behavioral: REACH-VIETNAM — Family caregiver education, stress-reduction, and skill-training related to providing care for a person with Alzheimer's disease
  Arms: REACH-VN

SUMMARY:
This is a cluster randomized controlled trial to determine the feasibility and preliminary effectiveness of culturally adapted psychosocial intervention for Alzheimer's family caregivers in Vietnam. The psychosocial intervention is being compared with an enhance control condition.

ELIGIBILITY:
Inclusion Criteria:

* Family member providing care to someone in household with Alzheimer's disease or a related dementia

Exclusion Criteria:

* Cognitively impaired

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-06-10 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ladson Hinton, MD, Principal Investigator — UC Davis
Locations (1):
- Vietnam National Geriatric Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Nguyen TA, Nguyen H, Pham T, Nguyen TH, Hinton L. A cluster randomized controlled trial to test the feasibility and preliminary effectiveness of a family dementia caregiver intervention in Vietnam: The REACH VN study protocol. Medicine (Baltimore). 2018 Oct;97(42):e12553. doi: 10.1097/MD.0000000000012553. PMID 30334942

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | REACH-VN | Enhanced Control
Started | 30 | 30
Completed | 25 | 26
Not Completed | 5 | 4
Not completed — caregiver demented, care recipient died | 3 | 3
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | REACH-VN | Enhanced Control | Total
Number analyzed (Participants) | 25 | 26 | 51
Age, Categorical [Count of Participants; unit: Participants] — Population: Data inadvertently not collected for two subjects.
  Participants
    number analyzed (Participants) | 25 | 24 | 49
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 17 | 15 | 32
    >=65 years | 8 | 9 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Data inadvertently not collected for two subjects.
  years
    number analyzed (Participants) | 25 | 24 | 49
    (all) | 59 (10.4) | 58.7 (13.9) | 58.8 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 21 | 44
  Male | 2 | 5 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 25 | 26 | 51
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 25 | 26 | 51
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Vietnam | 25 | 26 | 51
Zarit Burden Inventory - 4 item [Mean (Standard Deviation); unit: units on a scale] | 6.7 (2.1) | 6.8 (2.3) | 6.7 (2.2)

OUTCOME MEASURES:

1. Primary Outcome: Zarit Burden Inventory-4
Description: Measure of caregiver burden. Range is 0-16. Higher score indicates worse outcome (i.e., more burden).
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | REACH-VN | Enhanced Control
Number analyzed (Participants) | 25 | 26
score on a scale | 2.9 (2.4) | 5.5 (3.4)

2. Secondary Outcome: Patient Health Questionnaire-4
Description: Depressive and anxiety symptoms. Range is 0-12. Higher score indicates worse outcome (i.e., greater symptom severity).
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | REACH-VN | Enhanced Control
Number analyzed (Participants) | 25 | 26
units on a scale | 0.9 (1.0) | 2.9 (2.8)

3. Secondary Outcome: Alzheimer's Disease Knowledge Scale
Description: Scale that assess knowledge of Alzheimer's disease. Range is 0-30. Higher score is better outcome (i.e., more accurate knowledge).
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | REACH-VN | Enhanced Control
Number analyzed (Participants) | 25 | 26
score on a scale | 19.9 (3.2) | 20.1 (2.0)

ADVERSE EVENTS:
Time Frame: For each participant adverse events were collected for the duration of participation in the study (i.e., up to 3 months)
Arm/Group | REACH-VN | Enhanced Control
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Informed Consent Form (2018-04-02): https://cdn.clinicaltrials.gov/large-docs/74/NCT03587974/ICF_000.pdf
  • Statistical Analysis Plan (2020-03-01): https://cdn.clinicaltrials.gov/large-docs/74/NCT03587974/SAP_001.pdf
  • Study Protocol (2018-04-02): https://cdn.clinicaltrials.gov/large-docs/74/NCT03587974/Prot_002.pdf